CLINICAL TRIAL: NCT06960213
Title: STOP-HAE: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of siRNA Targeting of Prekallikrein With ADX-324 in Participants With Hereditary Angioedema
Brief Title: STOP-HAE: A Phase 3 Study of ADX-324 in HAE
Acronym: STOP-HAE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ADARx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-324-301
Record Dates: First submitted 2025-04-07; First posted 2025-05-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Angioedema; HAE; Hereditary Angioedema - Type 1; Hereditary Angioedema - Type 2
Keywords: HAE; Hereditary angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — RNA, Small Interfering; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ADX-324 Dose Level 1 (Experimental)
  Interventions: Drug: ADX-324
- ADX-324 Dose Level 2 (Experimental)
  Interventions: Drug: ADX-324
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-324 — siRNA duplex oligonucleotide
  Other Names: siRNA
  Arms: ADX-324 Dose Level 1; ADX-324 Dose Level 2
Drug: Placebo — saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Evaluate the efficacy safety, pharmacokinetics (PK), pharmacodynamics (PD), and health-related quality of life (HRQoL) measures in participants with Type I and Type II HAE.

DETAILED DESCRIPTION:
This Phase 3 study will evaluate the efficacy of 2 doses and regimens of ADX-324 in preventing HAE attacks compared with placebo in participants with Type I and Type II HAE. The study will also evaluate safety, pharmacokinetics (PK), pharmacodynamics (PD), and health-related quality of life (HRQoL) measures.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥18 years at the time of signing informed consent.
* Have a documented diagnosis of HAE-1/HAE-2 (Type I or II)
* Experience ≥1 Investigator-confirmed HAE attack in the first 4 weeks of Screening or ≥2 Investigator-confirmed HAE attacks in 8 weeks of Screening.
* Have access to, and the ability to use, at least one acute HAE therapy to treat HAE attacks (eg, plasma-derived or recombinant C1-INH concentrate or a BK2-receptor antagonist) that has previously been shown to be effective for the participant.
* Participants must be deemed medically appropriate for on-demand treatment as the sole medicinal management for their HAE during the study, per Investigator.
* Women of childbearing potential must have a negative serum pregnancy test during Screening and a negative urine pregnancy test on Study Day 1 before study drug administration and must agree to use acceptable contraceptive methods if engaged in sexual activity of childbearing potential (refer to Section 13.2.2) from the time of signing the informed consent form (ICF) until the EOS Visit or 1 month after study drug administration, whichever is longer.

Key Exclusion Criteria:

* Concurrent diagnosis of another form of recurrent angioedema. Examples include, but are not limited to, acquired angioedema, HAE with normal C1-INH (previously known as HAE Type III), idiopathic angioedema, and recurrent angioedema associated with urticaria.
* Any clinically significant medical history including, but not limited to, uncontrolled hypertension (defined as systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥ 100 mmHg despite therapy), uncontrolled diabetes mellitus (HbA1c >9.0%), or current cardiovascular disease, including recent acute coronary syndrome (within the past 6 months), congestive heart failure (NYHA Class III or IV), and significant arrhythmias.
* Any clinically significant renal disease
* Any clinically significant hepatic disease
* Exposure to any of the following LTP for HAE:

  1. Chronic prophylaxis with C1-INH (CINRYZE, HAEGARDA, RUCONEST) within 2 weeks prior to Screening.
  2. Chronic prophylaxis with berotralstat (ORLADEYO) within 3 weeks prior to Screening.
  3. Chronic prophylaxis with lanadelumab (TAKHZYRO) within 8 weeks prior to the Screening.
  4. Androgen use within 12 weeks prior to Screening.
* Received prior treatment with any RNA/DNA-based therapy for HAE (including ADX-324) or is intolerant of any prior RNA/DNA-based therapy for any condition, excluding vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of ADX-324 in preventing HAE attacks | Day 22 to Week 25
  The time-normalized number of Investigator-confirmed HAE attacks per month for ADX-324 Dose Level 1 vs placebo

SECONDARY OUTCOMES:
Efficacy of ADX-324 in preventing HAE attacks | Day 22 to Week 25
  The time-normalized number of Investigator-confirmed HAE attacks per month for ADX-324 Dose Level 2 vs placebo
Evaluate the effects of ADX-324 on the quality and pattern of HAE attacks | Day 22 to Week 25
  The time-normalized number of Investigator-confirmed HAE attacks requiring acute HAE therapy per month for ADX-324 vs placebo.
Evaluate the effects of ADX-324 on the quality and pattern of HAE attacks | Day 22 to Week 25
  The time-normalized number of moderate or severe Investigator confirmed HAE attacks per month for ADX 324 vs placebo.
Evaluate the effects of ADX-324 on the quality and pattern of HAE attacks | Day 22 to Week 25
  The proportion of participants who have not experienced an Investigator-confirmed HAE attack (HAE attack-free) for ADX 324 vs placebo.
Evaluate the effects of ADX-324 on the quality and pattern of HAE attacks | Day 22 to Week 25
  The proportion of participants with a clinical response defined as a ≥50%, ≥70%, or ≥90% reduction from baseline in Investigator-confirmed HAE attack rate for ADX 324 vs placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Masako Murai, MD, Study Director — ADARx Pharmaceuticals, Inc.
Locations (14):
- United States (10):
  - ADARx Clinical Site, Little Rock, Arkansas
  - ADARx Clinical Site, Walnut Creek, California
  - ADARx Clinical Site, Wheaton, Maryland
  - ADARx Clinical Site, Detroit, Michigan
  - ADARx Clinical Site, St Louis, Missouri
  - ADARx Clinical Site, Las Vegas, Nevada
  - ADARx Clinical Site, New York, New York
  - ADARx Clinical Site, Cincinnati, Ohio
  - ADARx Clinical Site, Columbus, Ohio
  - ADARx Clinical Site, Toledo, Ohio
- ADARx Clinical Site, Ottawa, Ontario, Canada
- ADARx Clinical Site, Hradec Králové, Czechia
- ADARx Clinical Site, Budapest, Hungary
- ADARx Clinical Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided